CLINICAL TRIAL: NCT06522100
Title: Use of Glucocorticoids Therapy in Acute Myocarditis With Severe Left Ventricular Dysfunction: a Multicenter Randomized Controlled Trial
Brief Title: Corticoid Therapy in Acute Myocarditis
Acronym: COTAM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP230855
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Myocarditis
Keywords: Acute myocarditis; Corticoids; Left ventricular dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, randomized, placebo controlled, superiority, double blinded trial with 2 parallel groups randomized in a 1:1 ratio.
  Patients will be hospitalized in Cardiology or Intensive Care Unit for a suspicion of an acute myocarditis. They will have an 2D-TTE to confirm a left ventricular dysfunction (LVEF < 50% and/or Global longitudinal strain [GLS] < -16%) and a cardiac magnetic resonance imaging or an endomyocardial biopsy will be performed to prove acute myocarditis. Coronary artery disease will be excluded by coronary angiography or Cardiac CT Scan. Once diagnosis of complicated AM with left ventricular dysfunction done, investigators will have 48 hours to include the patients and randomize them. They will benefit of placebo or experimental treatment in addition of conventional treatment for 6 months. At M6, end of participation for each patients, they will benefit of cardiologist consultation with TTE and cardiac magnetic resonance imaging.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Randomization in experimental group in addition to conventional HF therapy for 6 months.
  Interventions: Drug: Intravenous administration of Methylprednisolone; Drug: Oral Prednisone
- Control group (Placebo Comparator): Randomization in control group in addition to conventional HF therapy for 6 months.
  Interventions: Drug: Perfusion of placebo; Drug: Oral Prednisone placebo

INTERVENTIONS:
Drug: Intravenous administration of Methylprednisolone — Patients will take intravenous administration of Methylprednisolone (500mg/100ml by IV over 30 minutes per day) for 3 days.
  Arms: Experimental group
Drug: Oral Prednisone — After intravenous administration of Methylprednisolone patients will take by oral Prednisone 1mg/kg per day once a day (with a maximum dose of 90 mg per day for patients weighing > 90kg) for 1 month, followed with a progressive decrease of 10 mg Prednisone every 15 days until a dose of 10mg per day during 15 days (= stop).
  Arms: Experimental group
Drug: Perfusion of placebo — Patients will take perfusion of placebo (G5%: 100ml over 30 minutes per day) for 3 days.
  Arms: Control group
Drug: Oral Prednisone placebo — After the perfusion of placebo, patients will take by oral Prednisone placebo once a day for the same duration as that required if the patient was in the investigational medicinal products group (1 month + progressive decrease).
  Arms: Control group

SUMMARY:
Refer to the "Detailed Description" section.

DETAILED DESCRIPTION:
Introduction: Acute myocarditis (AM) is an inflammatory disease of the heart. The incidence is approximately 22 out of 100 000 patients annually. Clinically, it ranges from subclinical pauci-symptomatic forms to life-threatening arrhythmias, cardiogenic shock and sudden cardiac death. In approximately more than 70% of cases, AM resolves spontaneously. In the remaining patients, it evolves to a poor prognosis with left ventricular dilatation, reduced cardiac contractility and progression to chronic heart failure.

Complicated AM is defined as an AM with Left Ventricular Ejection Fraction (LVEF) < 50% and/or a sustained ventricular arrhythmia and/or a hemodynamic instability. Complicated AM is often associated with a poor prognosis (in example risk of heart transplantation of 10.4% at 30 days and 14.7% at 5-year follow up) whereas uncomplicated AM have none.

Administration of immunosuppressive treatment (IT) is still debated. According to experts' consensus, immunosuppressive treatment should be considered in complicated AM and should be used in recommended in case of fulminant myocarditis (acute myocarditis with a presentation of cardiogenic shock, ventricular arrhythmias, or multiorgan system failure). Nevertheless, there is no data on use of glucocorticoids (GC) in complicated AM.

Early application of high dose of GC in AM can control the cytokine storm and the inflammatory response, rather than suppressing the overall immune response. Best timing for their administration remains unknown. The aim of this multicenter controlled randomized study is to demonstrate the benefit of high dose of GC therapy on mortality and cardiac events in patients with AM and left ventricular (LV) dysfunction.

Hypothesis/Objective: The main objective is to evaluate in patients with acute myocarditis with left-ventricular dysfunction the efficacy of a pulse of Methylprednisolone IV for 3 days at diagnosis followed by Prednisone per os versus placebo IV followed by placebo per os in association with conventional Heart Failure (HF) therapy on the occurrence of Major Cardiovascular Events (MACE) and/or persistence of left ventricular dysfunction defined as LVEF < 50% and/or Global Longitudinal Strain (GLS) < -16% between baseline and at 6 months.

The primary endpoint is the Major Cardiovascular Events (MACE) and/or persistence of left ventricular dysfunction defined as LVEF < 50% and/or Global Longitudinal Strain (GLS) < - 16% between baseline (D-2) and 6 months (M6) follow up. MACE is a combined criterion that includes all-cause mortality, heart failure hospitalization, sustained ventricular arrhythmia, heart transplantation or assistance and recurrent acute myocarditis with LV dysfunction at 6 months.

Method: Phase III, prospective, randomized, placebo controlled, superiority, double blinded trial with 2 parallel groups randomized in a 1:1 ratio:

* Experimental group: Methylprednisolone IV for 3 days followed by Prednisone per os + conventional HF treatment.
* Control group: placebo of Methylprednisolone IV followed by placebo of Prednisone per os + conventional HF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written signed informed consent
* Affiliation to the French health care system or to another social protection scheme with the exception of State Medical Aid
* Active myocarditis defined by (all items are required):

  * Acute chest pain and/or unexplained heart failure and/or syncope and/or sustained ventricular arrhythmias and/or aborted sudden death and/or cardiogenic shock and/or ECG modification (atrioventricular block or bundle branch block or sinus arrest or ST or T waves change or ventricular arrhythmia or atrial fibrillation or abnormal Q waves)
  * And troponin rise (1,5 times the normal range)
  * And diagnosis of active myocarditis on Cardiac Magnetic Resonance (according to Lake-Louise criteria) or by histological evidence on endomyocardial biopsy (Dallas's criteria)
* Left-ventricular dysfunction defined as LVEF < 50% and/or GLS < -16% assessed with 2D-TTE
* Normal coronary angiography or CT Scan (without stenosis > 50%) during the previous year

Exclusion Criteria:

* Active coronary disease
* Other causes of chronic heart failure (coronary artery disease, primary valvular heart disease, congenital heart disease)
* Other etiology of myocarditis requiring corticosteroids treatment as giant cells myocarditis, eosinophilic myocarditis and cardiac sarcoidosis or immune checkpoint inhibitor myocarditis
* Other auto-immune or inflammatory disease requiring corticosteroids treatment within 6 months before enrolment
* Pregnancy or breastfeeding
* Woman of childbearing potential without effective method of birth control (included contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices)
* Patient deprived of liberty or under Curatorship/Tutorship, safeguard of justice, according to French law
* Foreseeable inability, according to the investigator, to participate in all the visits, treatments and measures provided for in the protocol
* Patient not speaking or understanding French
* Concomitant participation in another clinical trial on medical product for human use, to a clinical investigation on a medical device, to interventional study involving human participants or in the exclusion period at the end of a previous clinical trial on medical product for human use, a clinical investigation on a medical device, or study involving human participants. Participation in non-interventional research is permitted.
* Any medical and/or cognitive condition which limits the ability of participant to participate in study
* Contra-indication linked to steroids (Methylprednisolone and Prednisone) according to summary of product characteristics:

  * Any infectious condition excluding the specified therapeutic indications of Methylprednisolone and Prednisone
  * Certain evolving viruses (notably hepatitis, herpes, chickenpox, shingles)
  * Psychotic states not yet controlled by treatment
  * Recent live vaccines or live attenuated vaccines in patients receiving dosages greater than 20 mg/day of prednisone equivalent for more than two weeks and during the 3 months following the cessation of corticosteroid therapy (risk of generalized vaccine disease possibly fatal)
  * Hypersensitivity to the active substances or to any of the excipients
* Contra-indication linked to auxiliary drugs according to respective summary of product characteristics:

  * Beta-blockade
  * Angiotensin-converting-enzyme inhibitor (ACE-I)
  * Angiotensin receptor blockers (ARB)
  * Mineralocorticoid antagonists (MRA)
  * Angiotensin receptor-neprilysin inhibitor (ARNi)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-08-16 (Estimated); Study Completion 2028-08-16 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatments | 6 months
  Major Cardiovascular Events (MACE) and/or persistence of left ventricular dysfunction defined as LVEF < 50% and/or Global Longitudinal Strain (GLS) < - 16%. MACE is a combined criterion that includes all-cause mortality, heart failure hospitalization, sustained ventricular arrhythmia, heart transplantation or assistance and recurrent acute myocarditis with LV dysfunction.

SECONDARY OUTCOMES:
Changes in LVEF ≥ 50% | 6 months
  Changes in LVEF ≥ 50% at 6 months using 2D trans-thoracic echocardiography (2D-TTE)
Global Longitudinal Strain (GLS) ≥ -16% | 6 months
  Changes in Global Longitudinal Strain (GLS) ≥ -16% at 6 months using 2D-TTE
All-cause mortality | 6 months
  Occurred of a death
Heart failure hospitalization | 6 months
  Occurred of hospitalization for heart failure
Sustained ventricular arrhythmia | 6 months
  Occurred of sustained ventricular arrhythmia
Heart transplantation | 6 months
  Occurred of heart transplantation
Heart assistance by extracorporeal membrane oxygenation (ECMO), Intra-aortic balloon pump (IABP), Impella® device or Left Ventricular Assistance Devices (LVAD) | 6 months
  Need for heart assistance by extracorporeal membrane oxygenation (ECMO), Intra-aortic balloon pump (IABP), Impella® device or Left Ventricular Assistance Devices (LVAD)
Recurrence of acute myocarditis with LV dysfunction | 6 months
  Time to recurrence of acute myocarditis with LV dysfunction
Safety of the treatment regimens | 6 months
  Adverse events and serious adverse events
Adherence to the treatment regimen | 6 months
  Compliance to the treatment (premature ending of the treatment or proportion of non-administered doses of the treatment)
Evaluate quality of life using Minnesota living with heart failure questionnaire (MLHFQ) | 6 months
  Increased quality of life evaluated by Minnesota living with heart failure questionnaire during follow up. 21 questions rated from 0 to 5. Overall score from 0 to 105. The score increase with the adverse impact of heart failure.

IPD SHARING:
Plan to Share IPD: No
Datas are own by assistance publique - hopitaux de paris, please contact sponsor for further information.